CLINICAL TRIAL: NCT06653491
Title: Immediate Effects of the HVLA Talocrural Distraction Technique in Dorsiflexion, the Plantar Center of Pressure and the Percentage of Rearfoot Loading in Soccer Players
Brief Title: Immediate Effects of the HVLA Talocrural Distraction Technique in Soccer Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Professor of Department of Radiology, Rehabilitation and Physiotherapy, Faculty of Nursing, Physiotherapy and Podiatry, Universidad Complutense de Madrid, Madrid, Spain, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UComplutenseMadrid HVLA ankle
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Ankle Injury; Plantar Pressure
Keywords: ankle; manual therapy; plantar pressure center; mobility
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): high-speed, low-amplitude talocrural decompression technique and changes at the level of mobility and plantar pressure
  Interventions: Other: high-speed, low-amplitude talocrural decompression technique and changes at the level of mobility and plantar pressure
- Active Comparator (Active Comparator): simulated ankle technique and changes at the level of mobility and plantar pressure
  Interventions: Other: simulated ankle technique

INTERVENTIONS:
Other: high-speed, low-amplitude talocrural decompression technique and changes at the level of mobility and plantar pressure — high-speed, low-amplitude talocrural decompression technique and changes at the level of mobility and plantar pressure in a supine position
  Arms: Experimental
Other: simulated ankle technique — simulated ankle technique in a supine position
  Arms: Active Comparator

SUMMARY:
This clinical trial aims to evaluate the effect of a high-speed, low-amplitude physiotherapy technique at the ankle level, when performed on amateur soccer players.

DETAILED DESCRIPTION:
In this randomized, single-blind, cross-sectional and prospective clinical trial, the effect on ankle mobility and changes in plantar pressure centers obtained after performing a high-velocity, low-amplitude physiotherapy technique in amateur soccers will be assessed.

Two intervention groups are used; in one of them this treatment will be applied in a real way, and in the other one a simulation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years old
* Men that played or have played soccer as an amateur or professional on a regular basis
* No previous musculoskeletal history that would contraindicate HLVA techniques (recent fractures, osteosynthesis material placed in the joint, infections...)

Exclusion Criteria:

* Subjects under 18 years old
* Subjects who have suffered musculoskeletal pathology in the lower limb that contraindicates manipulation or who have a medical diagnosis of chronic ankle instability
* Subjects who suffer neurological or cognitive alterations that prevent the understanding of questionnaires or physical tests; and those who have not signed the informed consent documents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men that played or have played soccer as an amateur or professional on a regular basis
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Ankle range of motion | one day
  ankle dorsiflexion mobility with a manual dorsiflexion mobility test
plantar pressure centers | one day
  plantar pressure centers using stabilometric platform

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamali F, Sinaei E, Bahadorian S. The immediate effect of talocrural joint manipulation on functional performance of 15-40 years old athletes with chronic ankle instability: A double-blind randomized clinical trial. J Bodyw Mov Ther. 2017 Oct;21(4):830-834. doi: 10.1016/j.jbmt.2017.01.010. Epub 2017 Jan 25. PMID 29037635
- [Result] Manoel LS, Xixirry MG, Soeira TP, Saad MC, Riberto M. Identification of Ankle Injury Risk Factors in Professional Soccer Players Through a Preseason Functional Assessment. Orthop J Sports Med. 2020 Jun 24;8(6):2325967120928434. doi: 10.1177/2325967120928434. eCollection 2020 Jun. PMID 32637431
- [Result] Knuckles AM, Torp DM, Hubbard-Turner T, Donovan L, Thomas AC. Multi-axis destabilisation device influences plantar pressure distribution in adults with chronic ankle instability. Sports Biomech. 2022 Apr;21(4):501-516. doi: 10.1080/14763141.2021.1896773. Epub 2021 Mar 28. PMID 33779500